CLINICAL TRIAL: NCT05712447
Title: Duchenne Muscular Dystrophy Video Assessment Registry
Acronym: ARISE
Status: Active, not recruiting | Type: Observational
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: Department of Defense Duchenne Muscular Dystrophy Research Program (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAS-CAS005-01
Record Dates: First submitted 2022-11-30; First posted 2023-02-03 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne; DMD; Remote video assessment
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ARISE is a prospective and longitudinal clinical study of individuals with Duchenne Muscular Dystrophy (DMD) aimed at creating a database of functional motor abilities in this population to support validation efforts of the Duchenne Video Assessment (DVA).

DETAILED DESCRIPTION:
ARISE is a longitudinal, observational study of individuals with Duchenne muscular dystrophy (DMD). The Duchenne Video Assessment (DVA) is a home-based clinical outcome assessment that measures ease of movement through identification of compensatory movement patterns. The DVA directs caregivers to video record patients doing specific movement activities at home using a secure mobile application. In this study, participants will remotely complete the DVA in addition to existing DMD functional assessments (North Star Ambulatory Assessment (NSAA) and Performance of Upper Limb (PUL 2.0)) to evaluate the longitudinal measurement properties of the DVA.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 years of age at time of consent
* Written consent (English only) by adult participant or parent/legal guardian of minor participant
* Written assent (English only) if minor participant is at least 7 years of age
* Documentation provided for the participant's diagnosis of DMD (i.e., genetic report, clinic note)

Exclusion Criteria:

Participants will be excluded if they are unable to use a hand to hold a pen, pick up pennies or drive a powerchair.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited for this study through referrals from collaborators and advocacy groups as well as through direct marketing via social media, email, phone, or other appropriate methods. Advocacy groups will assist with the facilitation of recruitment by making recruitment materials available to the Duchenne community. Participants who provided consent to be contacted by Casimir staff for future studies and shared their contact information with Casimir staff may be contacted. Potential participants may also share their contact information directly with Casimir study staff to learn about the study. Additionally, recruitment for the study may also occur through postings with patient advocacy groups and on social media. Casimir will supply the advocacy groups with language for website postings and group emails.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Duchenne Video Assessment (DVA) | 24 months
  The DVA is a home-based clinical outcome assessment that measures ease of movement through identification of compensatory movement patterns. The DVA includes 18 standardized movement tasks that are assigned to participants based on functional subgroup. The DVA directs and trains caregivers to video record patients doing specific movement tasks at home using a secure mobile application. DVA videos are scored by DVA-certified physical therapists using validated scorecards with prespecified compensatory movement criteria.

SECONDARY OUTCOMES:
North Star Ambulatory Assessment (NSAA) | 24 months
  The NSAA is a 17-item tool used to measure functional motor abilities in ambulatory individuals with DMD. Physical therapists with experience administering the NSAA will remotely administer and record the live NSAA sessions via a secure video conference platform. Participants will receive the appropriate standardized testing equipment.
Performance of Upper Limb 2.0 (PUL 2.0) | 24 months
  The PUL 2.0 is a 22-item rating scale used to measure upper limb abilities in individuals with DMD. The test includes an entry test item to define starting functional level and 21 test items subdivided into shoulder level, elbow level, and distal level. Physical therapists with experience administering the PUL 2.0 will remotely administer and record the live PUL 2.0 sessions via secure video conference platform. Participants will receive the appropriate standardized testing equipment.
Caregiver Task-Specific Impression of Change | 24 months
  At each follow-up assessment timepoint, parents/legal guardians or recording partners will complete an electronic questionnaire to rate their impression of change in the participant's ability to perform each DVA movement task since the prior timepoint.

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Contesse, PhD, Principal Investigator — Emmes Endpoint Solutions
Locations (1):
- Emmes, Rockville, Maryland, United States